CLINICAL TRIAL: NCT02584465
Title: A Randomized, Open-label, Comparative, Multicenter, Phase II Study of the Efficacy and Safety of REGorafenib Versus Tamoxifen in Patients With Platinum-sensitive OVARian Carcinoma and Isolated Biological Progression
Brief Title: REGorafenib vsTamoxifen in Patients With Platinum-sensitive OVARian Carcinoma and Isolated Biological Progression
Acronym: REGOVAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ARCAGY/ GINECO GROUP (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GINECO-OV235
Record Dates: First submitted 2015-07-29; First posted 2015-10-22 (Estimated); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Ovarian Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Tamoxifen; regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A-Tamoxifen (Active Comparator): Tamoxifen 40mg/day 2 film-coated tablet containing 20 mg of Tamoxifen/day until progression
  Interventions: Drug: Tamoxifen
- B-Regorafenib (Experimental): Regorafenib 120mg/day 3 film-coated tablet containing 40 mg of Regorafenib/day, 3 weeks/4 until progression
  Interventions: Drug: Regorafenib

INTERVENTIONS:
Drug: Tamoxifen — Tamoxifen: 40 mg/day
  Arms: A-Tamoxifen
Drug: Regorafenib — Stivarga; 120mg/day
  Arms: B-Regorafenib

SUMMARY:
The objective of this randomized phase II is to evaluate the benefit of regorafenib for ovarian patients who reported a confirmed elevated CA-125 level under surveillance or bevacizumab, compared with tamoxifen.

DETAILED DESCRIPTION:
* After surgery, most of patients with advanced ovarian/primitive peritoneal /fallopian carcinoma received as first line treatment, carboplatin plus paclitaxel plus or minus bevacizumab for 6 cycles followed by surveillance or bevacizumab maintenance therapy up to one year (GOG (Burger et al.), ICON7 (Perren et al.), French national guidelines Saint Paul de Vence (www.arcagy.org)).
* This multi-modality approach achieves clinical responses in about 70% of patients, although a majority of women eventually relapse and die from disease progression. The first sign of relapse can be a progressively rising CA-125 (Tuxen et al.).
* Biochemical-recurrent of Epithelial Ovarian Cancer (EOC) is defined as CA-125 elevation above normal values without clinical evidence of disease, and can predate clinical disease by approximately 3-6 months (Tuxen et al.). Even if CA-125 elevation is a harbinger of EOC relapse, the question remains as to whether early therapeutic intervention can translate into extending the duration of survival.
* A few years ago, Rustin reported from ovarian cancer patients on surveillance after first line treatment with isolated elevated CA-125 (without RECIST/symptoms criteria) that there was no benefit to initiate a new chemotherapy compared to surveillance (Rustin et al. Lancet 2010; Rustin et al. Ann Oncol 2011).
* For patients under bevacizumab on maintenance phase at the time of the CA-125 elevation without RECIST or symptoms progression, data are scare. In the GOG0218 trial, elevated CA-125 did not totally complied with RECIST criteria progression. This study reported that the median PFS is longer in patients with continuous bevacizumab (14.1 months), compared to patients under placebo (10.3 months), using CA-125 & RECIST criteria, supporting the hypothesis that a maintenance treatment with an anti angiogenic agent allows delaying disease progression (Burger et al. N. Engl. J. Med. 2011). In an analysis of progression-free survival in which data for patients with increased CA-125 levels were censored, the median progression-free survival was 12.0 months in the control group but 18.0 months in the bevacizumab-throughout group (hazard ratio, 0.645; P<0.001). The relationship of CA-125 to progressive disease (PD) may be altered in bevacizumab (BV)-treated patients. In the Ocean trial elevated CA-125 was associated with forthcoming progression for the majority of the patients under bevacizumab (HR 0.48) in the platinum sensitive population (Aghajanian et al.).
* Current international recommendations are to continue the same strategy (surveillance or maintenance bevacizumab) until RECIST or symptomatic progression regardless of the CA-125 level.
* However, some can argue that a waiting attitude is deemed unacceptable due to patient anxiety over a rising CA-125 compelling a significant proportion of physicians to propose a therapeutic intervention, due to the nearness of the disease progression.
* Tamoxifen is an endocrine alternative treatment option in patients with rising CA-125. Hurteau et al. studies supported the use of tamoxifen showing a 17% response rate in measurable recurrent disease, 13% response rate in platinum resistant disease, observed stable disease in 38% of patients lasting a median of 3 months (Hatch, et al).
* The use of tamoxifen treatment as a control arm for isolated CA-125 is thus justified based on a favorable toxicity profile compared with available cytotoxic agents and the lack of interference with subsequent interventions beyond documentation of clinical progression (Marckman, et al). As patients have until today no benefit to introduce a new chemotherapy regimen for isolated elevated CA-125 (Rustin et al 2010), exploring new anti-angiogenic agent could be clinically relevant. Agents that inhibit tumor angiogenesis and invasion were considered to be ideal candidates for the experimental arm given their potential to prolong the duration of disease-free survival while exhibiting a more favorable toxicity profile than cytotoxic drugs.
* Pazopanib and other multi-kinase inhibitors such as cediranib, nintenanib reported activity in relapsing ovarian cancer (sensitive or resistant population) used alone in several phase II trials (Matulonis et al., Ledermann et al., and Friedlander et al.).
* Regorafenib is a new oral multi-kinase inhibitor. It inhibits kinases involved in angiogenesis (VEGFR 1-3, TIE 2), signaling in the tumor microenvironment (PDGFR-β, FGFR) and oncogenesis (KIT, RET and BRAF). Inhibition of tumor growth and formation of metastases were shown in vivo. Tumor activity has been reported in a variety of tumor types. Regorafenib is approved in Europe for the treatment of metastatic colorectal cancer in patients previously treated with, or who are not considered candidates for, available therapies. An application for GIST progressing after imatinib and sunitinib has obtained the AMM in Europe. The recommended dose is 160 mg taken once daily for 3 weeks followed by 1 week off therapy.

The objective of this randomized phase II is to evaluate the benefit of regorafenib for ovarian patients who reported a confirmed elevated CA-125 level under surveillance or bevacizumab, compared with tamoxifen.

ELIGIBILITY:
Main Inclusion Criteria:

I2 Histological confirmation of epithelial ovarian, fallopian tube, or primary peritoneal cancer, I3 Rising CA-125 (according to the Rustin/GCIG criteria, see appendix 10)) occurring more than 6 months after the last platinum-based chemotherapy cycle (platinum sensitive), I4 No symptom related to ovarian cancer progression, I6 1 or 2 prior lines of platinum-based chemotherapy followed either by surveillance or bevacizumab or olaparib (outside therapeutic trial) maintenance, I7 Before randomization, patients must be in CR, PR or SD (RECIST version 1.1) under surveillance or maintenance with bevacizumab or olaparib,

I8 Adequate bone marrow, liver and renal functions as assessed by the following laboratory tests conducted within 7 days before randomization:

* Absolute Neutrophil Count ≥ 1.5 G/L, platelets count ≥ 100 G/L, and hemoglobin ≥ 9g/dL,
* AST/ALT ≤ 3 x upper limit of normal (ULN) (or ≤ 5.0 x ULN if liver metastasis) and total bilirubin ≤ 1.5 x ULN, Alkaline phosphatase ≤ 2.5 x ULN
* Serum creatinine ≤ 1.5 x ULN,
* Glomerular filtration rate (GFR) ≥ 30 mL/min/1.73 m² according to the Modification of Diet Renal Disease (MDRD) abbreviated formula
* Lipase ≤ 1.5 x ULN
* Prothrombine time-international normalized ratio (PT-INR) < 1.5 x ULN. Patients who are therapeutically anticoagulated with an agent such as warfarin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in this parameter exists, I9 Women of childbearing potential and partners must agree to use adequate contraceptive method (if no previous bilateral annexectomies) during the whole study period and for up to 6 months after the last dose of study treatment; a negative pregnancy test must be obtained prior to randomization,

Main Exclusion Criteria:

E4 Past or concurrent history of neoplasm other than ovarian cancer, except for in situ carcinoma of the cervix uteri, in situ breast cancer and/or basal cell epithelioma. All treats and cures cancer more than 3 years before the study entry is allowed E5 Known history or symptomatic metastatic brain or meningeal tumors (head CT or MRI at screening to confirm the absence of central nervous system (CNS) disease if the patient has symptoms suggestive or consistent with progressive CNS disease), E6 Any prior radiotherapy to the pelvis or abdomen; surgery (including open biopsy) within 4 weeks before starting study drugs (24 hours for minor surgical procedures), or planned major surgery during the study treatment period, E7 Any prior treatment with anti angiogenic agent such as pazopanib, nintedanib or cediranib.

E8 Endocrine therapy administered within 3 years prior to randomization,

E13 History of any of the following :

* abdominal fistula,
* gastrointestinal perforation,
* intra-abdominal abscess,
* any malabsorption condition, E14 Clinically significant bleeding NCI-CTCAE version 4.3 Grade 3 or higher within 30 days before randomization, E15 Congestive heart failure New York Heart Association (NYHA) ≥ class 2, E17 Uncontrolled hypertension (systolic blood pressure (BP) > 150 mmHg or diastolic pressure > 90 mmHg despite optimal medical management), E21 Ongoing infection > Grade 2 according to NCI-CTCAE version 4.3. Hepatitis B is allowed if no active replication is present. Hepatitis C is allowed if no antiviral treatment is required, E23 Interstitial lung disease with ongoing signs and symptoms at the time of screening,

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2015-08-28 (Actual); Primary Completion 2021-09-19 (Actual); Study Completion 2021-09-19 (Actual)

PRIMARY OUTCOMES:
Progression Free survival (PFS) | 4 months
  PFS according to the RECIST 1.1 criteria, based on the investigator's assessment.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 4 months
Time to start of first subsequent chemotherapy (TFST) | 5 months
Second progression-Free Survival (PFS2) | 6 months
  PFS2 based on the investigator's assessment.
Overall Survival (OS) | 7 months
Adverse events | 7 months
  frequency of adverse events according to MedDRA terms

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Olivier, MD, Principal Investigator — olivier.tredan@lyon.unicancer.fr
Locations (21):
- France (21):
  - Hôpital Jean Minjoz, Besançon
  - Institut Bergonié, Bordeaux
  - Centre Hospitalier de Cholet, Cholet
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Oscar Lambret, Lille
  - Centre Hospitalier Universitaire Dupuytren, Limoges
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Hôpital de Mont-de-Marsan, Mont-de-Marsan
  - Centre Azuréen de Cancérologie, Mougins
  - ORACLE - Centre d'Oncologie de Gentilly, Nancy
  - Centre Catherine de Sienne, Nantes
  - Centre Hospitalier Régional d'Orléans, Orléans
  - Institut Mutualiste Montsouris, Paris
  - Clinique Francheville, Périgueux
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre CARIO - HPCA, Plérin
  - Centre Hospitalier Annecy Genevois, Pringy
  - Institut Jean Godinot, Reims
  - ICO Centre René Gauducheau, Saint-Herblain
  - Centre Hospitalier Universitaire Bretonneau, Tours